CLINICAL TRIAL: NCT01540669
Title: Dose-ranging Efficacy of 2-week Polydextrose Supplementation on Whole Gut Transit Time and Gastrointestinal Symptoms in Adults With Functional Constipation: A Double-blind, Randomized, Placebocontrolled Trial
Brief Title: Dose-Responsive Effect of Polydextrose on Whole Gut Transit Time
Acronym: PDX-Transit
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Danisco (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Q-PRE-0111-CLI-007
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Functional Constipation
Keywords: constipation; functional constipation; polydextrose; whole gut transit time
MeSH Terms: conditions — Constipation | interventions — polydextrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Polydextrose, low dose (Active Comparator): Polydextrose, low dose
  Interventions: Dietary Supplement: Polydextrose, low dose
- Polydextrose, medium dose (Active Comparator): Polydextrose, medium dose
  Interventions: Dietary Supplement: Polydextrose, medium dose
- Polydextrose, high dose (Active Comparator): Polydextrose, high dose
  Interventions: Dietary Supplement: Polydextrose, high dose
- Placebo powder (Placebo Comparator): Placebo powder
  Interventions: Dietary Supplement: Placebo powder

INTERVENTIONS:
Dietary Supplement: Polydextrose, low dose — 4g polydextrose powder will be mixed with beverage and consumed once per day for 2 weeks
  Arms: Polydextrose, low dose
Dietary Supplement: Polydextrose, medium dose — 8g polydextrose powder will be mixed with beverage and consumed once per day for 2 weeks
  Arms: Polydextrose, medium dose
Dietary Supplement: Polydextrose, high dose — 12g polydextrose powder will be mixed with beverage and consumed once per day for 2 weeks
  Arms: Polydextrose, high dose
Dietary Supplement: Placebo powder — Placebo powder will be mixed with beverage and consumed once per day for 2 weeks
  Arms: Placebo powder

SUMMARY:
The aim of the study is to test the effect of polydextrose on whole gut transit time and gastrointestinal symptoms in a dose-responsive manner.

DETAILED DESCRIPTION:
Given the promising, yet largely unsubstantiated, benefits of fiber supplementation, particularly polydextrose, on symptoms of functional constipation, the objective of this clinical trial is to evaluate the safety and effectiveness of 2-week supplementation of a proprietary polydextrose fiber product, in a dose-ranging fashion, on whole gut transit time and gastrointestinal symptoms in adults with functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Body mass index between 18.5 and 29.9 kg/m2 (encompasses normal weight and overweight)
* Meets the Rome III criteria for functional constipation as follows: (Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis):

Must meet 2 or more of the following criteria:

* Straining during at least 25% of defecations
* Lumpy or hard stools in at least 25% of defecations
* Sensation of incomplete evacuation for at least 25% of defecations
* Sensation of anorectal obstruction/blockage for at least 25% of defecations
* Manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor)
* Fewer than three defecations per week

  * Loose stools are rarely present without the use of laxatives
  * Insufficient criteria for irritable bowel syndrome
  * Ability of the participant (in the investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects
  * Consent to the study and willing to comply with study product and methods
  * Willingness to maintain a stable diet throughout the study
  * Consistent use and dose of chronic medication, if any, in the past 30 days

Exclusion Criteria:

* Major gastrointestinal complication (e.g. Crohn"s disease, colitis, celiac disease)
* Febrile diverticulitis within 1 year of screening
* Pelvic floor dysfunction
* Prior abdominal surgery that in the opinion of the investigator may present a risk for the subject or confound study results
* Prior abdominal surgery of the following type: gastric bypass, lap band, colectomy, removal of gall bladder
* Clinically significant underlying systemic illness that may preclude the subject"s ability to complete the trial or that may confound the study outcomes
* Any clinically relevant abnormalities in the physical examination or in laboratory variables before entry into the study
* Daily consumption of probiotics, prebiotics, fermented milk, and/or yogurt within 2 weeks of screening
* Laxative, fiber supplement, or other constipation medication (e.g. prokinetic drugs) use within 2 weeks of screening
* Antibiotic use within 1 month of enrollment
* Regular use of any drug or dietary supplement known to cause constipation (e.g. iron, opioids, sucralfate, misoprostol, 5-HT#- antagonists, antacids with magnesium or aluminum, or diarrhea medication)
* Anticipated major dietary or exercise changes during the study period
* Known allergies to any substance in the study product
* Pregnant or lactating female, or pregnancy planned during study period
* Eating disorder
* History of alcohol, drug, or medication abuse
* Participation in another study with any investigational product within 3 months of screening
* Investigator believes that the participant may be uncooperative and/or noncompliant and should therefore not participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Whole gut transit time | 2 weeks

SECONDARY OUTCOMES:
Patient assessment of constipation quality of life | 2 weeks
Patient assessment of constipation symptoms | 2 weeks
Bowel Function Index | 2 weeks
Adequate relief of constipation | 2 weeks
Bowel movement frequency | 2 weeks
Stool consistency | 2 weeks
Degree of straining | 2 weeks
Subjective assessment of bowel emptying | 2 weeks
Abdominal discomfort/bloating | 2 weeks
Overall product satisfaction | 2 weeks
Blood and urine safety analysis | 2 weeks
Adverse events | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Danese, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Terminated